CLINICAL TRIAL: NCT02426814
Title: Assessment of a Mobile Intervention to Increase Adherence to Asthma Medication Among Adolescents
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: CoheroHealth (Industry)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015_Spring_Sinai
Record Dates: First submitted 2015-04-07; First posted 2015-04-27 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Asthma
Keywords: Patient Compliance; Mobile Applications
MeSH Terms: conditions — Asthma; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Standard Care with Medication Monitoring (Sham Comparator): Patients will be given an inhaler sensor to monitor medication use and a sham version of the mobile app that will not include reminders or incentives.
  Intervention: inhaler sensor
  Interventions: Device: Inhaler sensor
- Medication Monitoring and Mobile App (Experimental): Patients will be given an inhaler sensor to monitor medication use and a mobile phone application with reminders to allow self-management of medication use.
  Interventions: inhaler sensor and mobile application for asthma adherence
  Interventions: Device: Inhaler sensor; Behavioral: Mobile application for asthma adherence

INTERVENTIONS:
Device: Inhaler sensor — Inhaler sensor strap that tracks inhaler use.
Behavioral: Mobile application for asthma adherence — Mobile phone application that sends reminders and allows patients to self-manage their medication adherence.
  Arms: Medication Monitoring and Mobile App

SUMMARY:
The purpose of this study is to assess the use of a mobile health intervention to improve adherence to asthma medication among adolescents. The intervention consists of an inhaler sensor strap to monitor asthma inhaler use and a mobile phone application to remind and incentivize patients to use their medication. This study will assess medication use throughout a 12 week study in patients who receive a mobile app with reminders, asthma control as measured by the ACT [asthma control test], and lung function as measured by spirometry.

ELIGIBILITY:
Inclusion Criteria:

* Age 11-19
* Asthma diagnosis
* Currently prescribed a hydrofluoroalkane (HFA) asthma controller medication
* English-speaking
* Has a smartphone or access to a smartphone or tablet

Exclusion Criteria:

* Pregnant
* Foster Care
* Emancipated minor

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Real-time medication adherence in patients using mobile app compared to standard care. | 12 weeks
  Analysis of real-time medication use data in the experimental [app + sensor] arm vs the sensor only arm.

SECONDARY OUTCOMES:
Asthma control in patients using mobile app compared to standard care | 12 weeks
  Analysis of the ACT [asthma control test] at baseline and follow up for patients in each arm to assess changes in asthma control with use of the mobile app.
Change in lung function with use of a mobile health tool for asthma adherence | 12 weeks
  Measure change in spirometry by comparing force expiratory volume at one second [FEV1] and forced vital capacity [FVC] at baseline and 12 week visit.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ting, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Michael Parides, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No